CLINICAL TRIAL: NCT07234721
Title: A Phase I Clinical Study of SL4903 Autologous T-Cell Injection for the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: SL4903 CAR-T Therapy for Relapsed/Refractory Multiple Myeloma
Acronym: SL4903
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025098
Record Dates: First submitted 2025-09-16; First posted 2025-11-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Relapsed and Refractory Multiple Myeloma (RRMM)
Keywords: BCMA+GPRC5D; SL4903; Multiple Myeloma; CART
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: ARM 1: dosage 1*10^6 CART cells/Kg; ARM 2: dosage 2*10^6 CART cells/Kg; ARM 3: dosage 3*10^6 CART cells/Kg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: dosage 1×10⁶ CAR⁺ cells/kg (Experimental): In this dosage cohort (1×10⁶ CAR⁺ cells/kg). A total of 3-6 subjects are expected to be enrolled to evaluate the safety and tolerability of SL4903 autologous T-cell injection and to determine the maximum tolerated dose (MTD).
  Dose-Escalation Rules
  • In the "3 + 3" phase, one subject is enrolled into each dose level and observed for 28 days after cell infusion (the observation period may be prolonged at the investigator's discretion).
  Interventions: Drug: SL4903 Autologous T-Cell Injection
- Arm 2: dosage 2×10⁶ CAR⁺ cells/kg (Experimental): In this dosage cohort (2×10⁶ CAR⁺ cells/kg). A total of 3-6 subjects are expected to be enrolled to evaluate the safety and tolerability of SL4903 autologous T-cell injection and to determine the maximum tolerated dose (MTD).
  Dose-Escalation Rules
  • In the "3 + 3" phase, one subject is enrolled into each dose level and observed for 28 days after cell infusion (the observation period may be prolonged at the investigator's discretion).
  Interventions: Drug: SL4903 Autologous T-Cell Injection
- Arm 3: dosage 3×10⁶ CAR⁺ cells/kg (Experimental): In this dosage cohort (3×10⁶ CAR⁺ cells/kg). A total of 3-6 subjects are expected to be enrolled to evaluate the safety and tolerability of SL4903 autologous T-cell injection and to determine the maximum tolerated dose (MTD).
  Dose-Escalation Rules
  • In the "3 + 3" phase, one subject is enrolled into each dose level and observed for 28 days after cell infusion (the observation period may be prolonged at the investigator's discretion).
  Interventions: Drug: SL4903 Autologous T-Cell Injection

INTERVENTIONS:
Drug: SL4903 Autologous T-Cell Injection — Eligible subjects, identified through application of inclusion/exclusion criteria, will be evaluated for tumor type, tumor burden, vital-sign status, and other comprehensive factors before receiving SL4903(1×10⁶ CAR⁺ cells/kg) cellular therapy.
  Arms: Arm 1: dosage 1×10⁶ CAR⁺ cells/kg
Drug: SL4903 Autologous T-Cell Injection — Eligible subjects, identified through application of inclusion/exclusion criteria, will be evaluated for tumor type, tumor burden, vital-sign status, and other comprehensive factors before receiving SL4903(2×10⁶ CAR⁺ cells/kg) cellular therapy.
  Arms: Arm 2: dosage 2×10⁶ CAR⁺ cells/kg
Drug: SL4903 Autologous T-Cell Injection — Eligible subjects, identified through application of inclusion/exclusion criteria, will be evaluated for tumor type, tumor burden, vital-sign status, and other comprehensive factors before receiving SL4903(3×10⁶ CAR⁺ cells/kg) cellular therapy.
  Arms: Arm 3: dosage 3×10⁶ CAR⁺ cells/kg

SUMMARY:
This is a Phase I, single-center, single-arm, open-label clinical study to evaluate the safety, tolerability, and preliminary efficacy of SL4903 autologous T-cell injection (CAR-T cell therapy) in adult patients with relapsed or refractory multiple myeloma (r/r MM) who have failed prior standard therapies.

The study employs a "3+3" dose-escalation design with three planned dose levels (1×10⁶, 2×10⁶, and 3×10⁶ CAR+ cells/kg). Approximately 9 to 18 evaluable subjects will be enrolled to determine the maximum tolerated dose (MTD) and recommended Phase II dose (RP2D), and to characterize the safety profile and potential anti-myeloma activity of SL4903.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet ALL of the following conditions:

1. Age 18-75 years; either sex.
2. Able to understand the study and provide voluntary written informed consent.
3. Histologically and/or cytologically confirmed multiple myeloma according to IMWG 2016 criteria, meeting the following conditions:

   1. Patients must have received at least one prior line of anti-myeloma therapy, including treatment with proteasome inhibitors (PIs), immunomodulatory drugs (IMiDs), and anti-CD38 monoclonal antibodies, or patients with multiple myeloma refractory to proteasome inhibitors, immunomodulatory drugs, and anti-CD38 monoclonal antibodies;
   2. Documented evidence of disease progression or failure to achieve complete response (CR) following the last line of therapy, as assessed by the investigator according to IMWG criteria.
4. Measurable disease at screening, defined as meeting one or more of the following criteria:

   * Serum M-protein ≥0.5 g/dL
   * Urinary M-protein ≥200 mg/24 h
   * Abnormal serum FLC ratio (<0.26 or >1.65) with involved FLC ≥10 mg/dL
   * Soft tissue extramedullary disease (EMD) identified by radiographic imaging with a longest diameter ≥ 2 cm
5. ECOG performance status 0-2.
6. Adequate organ function:

   1. Serum creatinine ≤150 µmol/L or calculated creatinine clearance (Cockcroft-Gault) ≥40 mL/min (may be relaxed for acute MM-related renal impairment at investigator discretion).
   2. Total bilirubin ≤2×ULN; ALT ≤3×ULN; AST ≤3×ULN.
   3. Normal diastolic function on echocardiography, LVEF ≥50 %, no significant arrhythmia.
   4. No active pulmonary infection; oxygen saturation on room air >90 %.
7. No contraindication to leukapheresis: Hemoglobin ≥ 60 g/L, platelets ≥ 50 × 10⁹/L, and lymphocytes ≥ 0.3 × 10⁹/L.
8. Life expectancy >12 weeks.
9. Women of child-bearing potential must have a negative urine pregnancy test and must not be breastfeeding; all men and women with reproductive potential must use effective contraception throughout the study.

Exclusion Criteria

A subject will be excluded if ANY of the following apply:

1. History of severe immediate hypersensitivity to any study drug.
2. Central nervous system (CNS) disorders such as epilepsy, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, or neuropathy (resolved cases without residual symptoms may be exempted at the investigator's discretion). Active CNS involvement, prior CNS myelomatous disease, or meningeal/spinal cord involvement signs must be excluded.
3. Prior traumatic brain injury, cerebrovascular accident, significant cerebral ischemia, or intracranial hemorrhage.
4. Concurrent uncontrolled malignancies other than adequately treated cervical carcinoma in situ, basal-cell or squamous-cell skin carcinoma, localized prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery, or thyroid cancer after curative surgery.
5. Clinically significant cardiovascular disease, e.g., uncontrolled or symptomatic arrhythmia, congestive heart failure, or NYHA class III/IV cardiac disease; myocardial infarction, coronary angioplasty/stenting, unstable angina, or other clinically relevant cardiac disorders within 12 months before enrollment.
6. Any severe comorbidity or condition judged by the investigator to increase subject risk or interfere with the study, including but not limited to liver cirrhosis or recent major trauma.
7. Prior BCMA- and/or GPRC5D-directed CAR-T therapy.
8. Allogeneic hematopoietic stem-cell transplantation within 6 months before screening, or any immunosuppressive therapy for graft-versus-host disease during screening.
9. Autoimmune disease, immunodeficiency, or need for immunosuppressants (except low-dose corticosteroids).
10. Uncontrolled active infection, including but not limited to active tuberculosis; suspected or proven uncontrolled fungal, bacterial, viral, or other infections.
11. Live attenuated vaccine within 4 weeks before leukapheresis.
12. Active hepatitis (HBV-DNA or HCV-RNA above the lower limit of detection), syphilis infection, congenital or acquired immunodeficiency including HIV, EBV or CMV viremia (DNA above the lower limit of detection).
13. History of alcohol abuse, drug abuse, or psychiatric illness.
14. Inability to meet the following washout requirements prior to PBMC collection:

    1. Corticosteroids: no more than 5 mg prednisone (or equivalent) within 72 h.
    2. Anti-tumor therapies: targeted therapy, epigenetic therapy, investigational drugs/devices-discontinued ≥14 days or ≥5 half-lives (whichever is longer); anti-myeloma monoclonal antibodies-≥21 days; cytotoxic therapy-≥14 days; proteasome inhibitors-≥14 days; immunomodulatory drugs-≥7 days.
    3. Radiotherapy: completed ≥4 weeks before leukapheresis, except if the radiation field covers ≤5 % of marrow reserves.
    4. Anti-T-cell antibodies (e.g., alemtuzumab): discontinued ≥8 weeks.
15. Any condition judged by the investigator to render the subject unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Number and incidence rate of adverse events following intravenous infusion of SL4903 cells | one month
  Within one month after cell infusion, all documented adverse events-including cytokine-release syndrome and neurotoxicity-will be analyzed for incidence, frequency, and severity to evaluate the safety of SL4903 and to determine the maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Overall response rate (ORR) | at 3, 6, 9, 12, 18, and 24-month after CAR-T infusion
  Percentage of subjects who achieved partial response (PR) or better according to IMWG Uniform Response Criteria for Multiple Myeloma
Complete response rate (CRR) | at 3, 6, 9, 12, 18, and 24-month after CAR-T infusion
  Percentage of subjects who achieved complete response (CR) or stringent complete response (sCR) according to IMWG Uniform Response Criteria for Multiple Myeloma
Time to Response (TTR) | Minimum of 2 years post SL4903 CAR-T infusion
  Time from SL4903 CAR-T infusion to first documentation of response evaluated by investigators
Progression-free Survival (PFS) | Minimum of 2 years post SL4903 CAR-T infusion
  Time from SL4903 CAR-T infusion to first documentation of progressive disease (PD), or death due to any cause, whichever occurs first
Duration of Response (DOR) | Minimum of 2 years post SL4903 CAR-T infusion
  Time from first response evaluated by investigators to disease progression or death from any cause
Overall Survival (OS) | Minimum of 2 years post SL4903 CAR-T infusion
  Time from SL4903 CAR-T infusion to time of death due to any cause
Minimal Residual Disease (MRD) negative rate | at 3, 6, 9, 12, 18, and 24-month after CAR-T infusion
  Proportion of subjects who achieved MRD negative
Pharmacokinetic (Cmax) | at day0 to day28 after CAR-T infusion
  Testing CARgene copies and CAR-T/T% in peripheral blood by qPCR and Flow cytometry，then analysising the Cmax.
Pharmacokinetic (Tmax) | at day0 to day28 after CAR-T infusion
  Testing CARgene copies and CAR-T/T% in peripheral blood by qPCR and Flow cytometry，then analysising the time to peak (Tmax).
Pharmacokinetic (AUCday0~28) | at day0 to day28 after CAR-T infusion
  Testing CARgene copies and CAR-T/T% in peripheral blood by qPCR and Flow cytometry，then analysising the AUC(day0~28).
proportion of peripheral plasma cells | at day0 , day7, day10, day14 and day28 after CAR-T infusion
  The proportion of peripheral plasma cells at various time points
cytokines level | at day0 , day7, day10, day14 and day28 after CAR-T infusion
  The release amount of cytokines at various time points

CONTACTS AND LOCATIONS:
Overall Officials: An, Principal Investigator — Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences,Tianjin

IPD SHARING:
Plan to Share IPD: No